CLINICAL TRIAL: NCT02876796
Title: A Randomized, Double-Blind, Placebo-Controlled Study To Evaluate the Pharmacodynamic Effects of A Single Oral Dose of NDI-010976 in Healthy Adult Subjects
Brief Title: Study to Evaluate the Pharmacodynamic Effects of a Single Oral Dose of GS-0976 (NDI-010976) in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Nimbus Apollo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 0976-103
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: PD Effects of GS-0976 (NDI-010976) on Fractional DNL
Keywords: fractional de novo lipogenesis; DNL; pharmacodynamic; pharmacokinetic
MeSH Terms: interventions — firsocostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 50 mg GS-0976 (Cohort 1) (Experimental): Sequence 1:
  Period 1 (2 days): 50 mg (1 x 50 mg capsule) + IV infusion 1-13C acetate and fructose solution; Washout Period (minimum of 5 days); Period 2 (2 days): placebo + IV infusion 1-13C acetate and fructose solution
  Sequence 2:
  Period 1 (2 days): placebo + IV infusion 1-13C acetate and fructose solution; Washout Period (minimum of 5 days); Period 2 (2 days): 50 mg (1 x 50 mg capsule) + IV infusion 1-13C acetate and fructose solution
  Interventions: Drug: GS-0976; Drug: Placebo; Other: 1-13C acetate; Other: Fructose solution
- 200 mg GS-0976 (Cohort 2) (Experimental): Sequence 3:
  Period 1 (2 days): 200 mg (1 x 200 mg capsule) + IV infusion 1-13C acetate and fructose solution; Washout Period (minimum of 5 days); Period 2 (2 days): placebo + IV infusion 1-13C acetate and fructose solution
  Sequence 4:
  Period 1 (2 days): placebo + IV infusion 1-13C acetate and fructose solution; Washout Period (minimum of 5 days); Period 2 (2 days): 200 mg (1 x 200 mg capsule) + IV infusion 1-13C acetate and fructose solution
  Interventions: Drug: GS-0976; Drug: Placebo; Other: 1-13C acetate; Other: Fructose solution
- 20 mg GS-0976 (Cohort 3) (Experimental): Sequence 5:
  Period 1 (2 days): 20 mg (2 X 10 mg capsule) + IV infusion 1-13C acetate and fructose solution; Washout Period (minimum of 5 days); Period 2 (2 days): placebo + IV infusion 1-13C acetate and fructose solution
  Sequence 6:
  Period 1 (2 days): placebo + IV infusion 1-13C acetate and fructose solution; Washout Period (minimum of 5 days); Period 2 (2 days): 20 mg (2 X 10 mg capsule) + IV infusion 1-13C acetate and fructose solution
  Interventions: Drug: GS-0976; Drug: Placebo; Other: 1-13C acetate; Other: Fructose solution

INTERVENTIONS:
Drug: GS-0976 — Capsule(s) administered orally
  Other Names: NDI-010976
Drug: Placebo — Capsule(s) administered orally
Other: 1-13C acetate — 10 g ± 0.25 g in 1000 mL 0.45% saline solution administered intravenously for 19 hours
Other: Fructose solution — Fructose solution administered orally under fasted conditions immediately after study drug and every 30 minutes for a total of 20 doses

SUMMARY:
The primary objective of this study is to assess the pharmacodynamic (PD) effects of GS-0976 (NDI-010976) on fractional de novo lipogenesis (DNL) following a single oral dose administration in overweight and/or obese, but otherwise healthy, male adults.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and/or obese, but otherwise healthy males
* Weight ≥ 50.0 kg
* Body Mass Index (BMI): 25.0 - 32.0 kg/m^2, inclusive

Exclusion Criteria:

* Intolerance to or malabsorption of fructose
* A history of clinically significant gastrointestinal disease and/or surgery, which would result in the subject's inability to absorb or metabolize the study drug (e.g., gastrectomy, gastric bypass, cholecystectomy).
* In the opinion of the Investigator, a history of clinically significant hematologic, renal, hepatic, bronchopulmonary, neurological, psychiatric, metabolic , endocrine disorder (e.g., diabetes, thyroid disease), or cardiovascular disease.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in fractional DNL (% new palmitate) | Predose and up to 10 hours postdose
Change in DNL over time following administration of GS-0976 and placebo | Predose and up to 10 hours postdose
Change from baseline over time in adiponectin | Baseline and up to 10 hours postdose
Percent change from baseline over time in adiponectin | Baseline and up to 10 hours postdose
Change from baseline over time in leptin | Baseline and up to 10 hours postdose
Percent change from baseline over time in leptin | Baseline and up to 10 hours postdose
Change from baseline over time in blood ketones | Baseline and up to 10 hours postdose
Percent change from baseline over time in blood ketones | Baseline and up to 10 hours postdose
Change from baseline over time in lipid profile | Baseline and up to 10 hours postdose
Percent change from baseline over time in lipid profile | Baseline and up to 10 hours postdose

SECONDARY OUTCOMES:
Number and severity of treatment-emergent adverse events (TEAEs) following single oral doses of GS-0976 and placebo | Up to 42 days
Percentage of participants experiencing abnormal clinical laboratory tests | Up to 42 days
Pharmacokinetics (PK) of GS-0976 and its metabolite: tmax | Baseline and up to 10 hours postdose
  Tmax is defined as the time (observed time point) of Cmax.
PK of GS-0976 and its metabolite: Cmax | Baseline and up to 10 hours postdose
  Cmax is defined as the maximum concentration of drug.
PK of GS-0976 and its metabolite: AUC_0-t | Baseline and up to 10 hours postdose
  AUC_0-t is defined as the concentration of drug over time from time zero to time "t".

CONTACTS AND LOCATIONS:
Overall Officials: Rob Myers, MD, Study Director — Gilead Sciences
Locations (1):
- Phoenix, Arizona, United States